CLINICAL TRIAL: NCT00491712
Title: Comparison of Efficacy Between Silicone Ahmed Glaucoma Valves With and Without Intravitreal Triamcinolone Injection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Federal University of São Paulo (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Glau00036
Record Dates: First submitted 2007-06-25; First posted 2007-06-26 (Estimated); Last update posted 2007-06-26 (Estimated); Status verified 2007-03

CONDITIONS: Neovascular Glaucoma
Keywords: Glaucoma; Neovascular Glaucoma; Drainage implant devices; Silicone Ahmed Tube; Triamcinolone
MeSH Terms: conditions — Glaucoma, Neovascular; Glaucoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Glaucoma drainage implant with/without triamcinolone

SUMMARY:
The management of neovascular glaucoma (NVG) is a challenge for the ophthalmologist and surgery is frequently needed to control IOP. The success rates of a drainage device is usually lower in NVG than in other forms of glaucoma. Triamcinolone intra-vitreous injections acetate has been used to treat macular edema secondary to diabetic retinopathy and central retinal vein occlusion and also to control inflammation in ophthalmologic surgeries.

In the present study we will compare the outcome and complications of Silicone Ahmed Valve in GNV eyes with and without intra-vitreous triamcinolone injection.

DETAILED DESCRIPTION:
The management of neovascular glaucoma (NVG) is a challenge for the ophthalmologist and surgery is frequently needed to control intraocular pressure (IOP). The success rates of a drainage device is usually lower in NVG than in other forms of glaucoma. Triamcinolone intra-vitreous injections acetate has been used to treat macular edema secondary to diabetic retinopathy and central retinal vein occlusion and also to control inflammation in ophthalmologic surgeries.

In the present study we will compare the outcome and complications of Silicone Ahmed Valve in GNV eyes with and without intra-vitreous triamcinolone injection.

49 Patients with clinically uncontrolled neovascular glaucoma were selected from the glaucoma sector of Federal university of Sao Paulo. After retinal panfotocoagulation (RPF), patients who still are uncontrolled are enrolled to the study. Patients were randomized to one of two groups:

1. Silicone Ahmed Implant
2. Silicone Ahmed Implant with intra-vitreous Triamcinolone injection

Inclusion Criteria:

Patients with NVG and uncontrolled IOP despite the use of maximum tolerated glaucoma medication Patients over 18 years old. Patients who can understand and sign the inform consent form.

Exclusion Criteria:

Active Sclerites Uveitic NVG Previous psiquiatric condition Patients who can understand and sign the inform consent form Visual acuity worse than hand motion Previous retina surgery with buckle implant

Surgery description A fornix-based conjunctival flap was created between two adjacent recti muscles. Before placement of the tube implant body to the sclera, tube was irrigated with saline solution to open the valve mechanism. The implant's polypropylene body was sutured to sclera with 6.0 silk suture. The tube then trimmed and the anterior chamber was entered from 1mm posterior to corneoscleral limbus with 23-gauge needle. A human donor scleral flap was placed over the tube and sutured to the sclera with 10.0 nylon suture. The conjunctiva was sutured to the limbus. In the triamcinolone group, a intra-vitreous injection of 0,1mL triamcinolone acetate (40mg/ml) was performed with a 30-gauge needle.

Follow up after surgery was in the 1st, 4th, 7th, 15th, 30th days and after that monthly or whenever needed for clinical reasons.

ELIGIBILITY:
Inclusion Criteria:

* Patients with NVG and uncontrolled IOP despite the use of maximum tolerated glaucoma medication
* Patients over 18 years old.
* Patients who can understand and sign the inform consent form.

Exclusion Criteria:

* Active Sclerites
* Uveitic Neovascular glaucoma
* Previous psiquiatric condition
* Patients who can understand and sign the inform consent form
* Visual acuity worse than hand motion
* Previous retina surgery with buckle implant

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2005-09; Study Completion 2007-06 (Estimated)

PRIMARY OUTCOMES:
intra ocular pressure after the surgery in both groups | monthly

SECONDARY OUTCOMES:
complication rates after surgery | monthly

CONTACTS AND LOCATIONS:
Overall Officials: Augusto Paranhos Jr, PHD, Principal Investigator — Federal University of São Paulo
Locations (1):
- Federal University of Sao Paulo, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Sivak-Callcott JA, O'Day DM, Gass JD, Tsai JC. Evidence-based recommendations for the diagnosis and treatment of neovascular glaucoma. Ophthalmology. 2001 Oct;108(10):1767-76; quiz1777, 1800. doi: 10.1016/s0161-6420(01)00775-8. PMID 11581047